CLINICAL TRIAL: NCT01020162
Title: Treatment of Ilioinguinal Entrapment Syndrome - a Randomised Controlled Trial
Brief Title: Treatment of Ilioinguinal Entrapment Syndrome - an Often Overlooked Cause of Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Lennart Hahn, MD PHD, Dept of Obstetrics&Gynecology, Sahlgrenska Academy at the University of Gothenburg
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 429-05
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Chronic Pelvic Pain
Keywords: Chronic pelvic pain; ilioinguinal nerve entrapment; randomized study; Chronic pelvic pain in women
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-surgical (Active Comparator): TENS, amitriptyline, gabapentin.
  Interventions: Drug: Amitryptiline, gabapentin
- Surgical intervention (Active Comparator): Resection of the ilioinguinal nerve
  Interventions: Procedure: Resection of the ilioinguinal nerve

INTERVENTIONS:
Drug: Amitryptiline, gabapentin — For amitryptiline starting dose 20-30 mg at night, increasing until clinical effect. For gabapentin was the initial dose 300 mg tid with rapid increases up to 800 mg tid.
  Other Names: Amitryptiline - Saroten; Gabapentin - Neurontin
  Arms: Non-surgical
Procedure: Resection of the ilioinguinal nerve — In general anaesthesia the nerve was identified and resected as central as possible
  Arms: Surgical intervention

SUMMARY:
Neuralgic pain caused by entrapment of peripheral nerves is an often overlooked cause of chronic pelvic pain. The objective of the present study was to assess pain and quality of life in women with pain caused by entrapment of the ilioinguinal nerve, iatrogenic after surgery but also found without previous surgery. In a controlled prospective cross-over study 19 women were randomized either to medical treatment or to resection of the nerve. Statistically significant improvements were found after surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Pelvic pain in which a careful investigation has shown signs of ilioinguinal nerve entrapment

Exclusion Criteria:

* Drug abuse

Ages: 15 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 1995-09; Primary Completion 2006-12 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Improvements in pain according to Visual Analogue Scales. Improvements in quality of life according to Psychological General Well-Being-scales. | At least one year after intervention,in some cases more then five years.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Milsom, MD,PhD, Study Chair — Dept Obstetrics&Gynecology, Sahlgrenska Academy at the University of Gothenburg, Sweden
Locations (1):
- Dept Obstetrics&Gynecology/East Hospital, Gothenburg, Sweden